CLINICAL TRIAL: NCT00362401
Title: Patients Perception of Mechanical Heart Valve Sounds: Psychoacoustics and Quality of Life
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Heart and Diabetes Center North Rhine-Westphalia (Other)
Responsible Party: University of Aarhus - Thais A. Pedersen, Thais A. Pedersen - University of Aarhus
Other Study IDs: 20050213; 20050213 - 19/04-2006
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Results first posted 2009-09-07 (Estimated); Last update posted 2009-09-07 (Estimated); Status verified 2009-08

CONDITIONS: Heart Valve Diseases
Keywords: Psychoacoustics; Quality of Life; Heart Valve Prosthesis
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the sound pressure levels (SPLs) from three of the most frequently implanted mechanical heart valve prostheses, in order to determine whether there was any significant difference between the intensities of the valve sounds

DETAILED DESCRIPTION:
Patient's perception of mechanical heart valve sounds: psychoacoustics and quality of life

Background: Approximately 90.000 mechanical prosthetic heart valves are implanted every year all over the world. They generate a clicking sound at closure, which can be a major problem for some patients. About 12% of them all experience annoyance, concentration disturbance, sleeping disorders and social embarrassment. All those factors could affect patients' quality of life.

Aim: to compare the sound pressure levels (SPLs) from three of the most frequently implanted mechanical heart valve prostheses, in order to determine whether there was any significant difference between the intensities of the valve sounds.

Material and Methods: We intended to include 150 patients with an implanted mechanical heart valve (ATS Medical, Medtronic-Hall or St. Jude Medical) in the aortic position between 3 months and 4 years before the analysis. For logistical reasons, the actual number of the patients included was 84. The total conducted valve sound was measured (by a method designed by the authors) for each patient. The measures took place in a bioacoustical laboratory built with a sound-insulated chamber with a very low background noise, designed for the purposes of the study. The measures were performed in German patients followed by "The Heart Centre" in Bad Oeynhausen (Herz- und Diabeteszentrum Nordrhein Westfalen, University of Bochum), where the mentioned laboratory is constructed. The sound analysis of the present study was conducted in a specially designed soundproof bioacoustic laboratory, which isolates the outside sound and vibration from the environment indoors. Inside the laboratory, heavy soundinsulated curtains were placed between the patient and the investigator chambers. The total background noise inside the patient chamber was 19 dB(A), and this was reduced further to 9 dB(A) by using a 250 Hz high-pass filter. The sounds were recorded with the patient in the supine position, and without clothes covering the chest. The valve closing sounds were recorded using a microphone (Brüel and Kjær 4179) placed 5 cm above the patient's chest. This sound was then preamplified (Brüel and Kjær 2660), amplified (Brüel and Kjær 2610) and 250 Hz high-pass filtered (Krohn-Hite 3944) (see Fig. 1). All valve sounds were recorded by the same experienced investigator and stored on an instrumentation recorder (TEAC 510) for later off-line analysis. The data acquisition time for each patient was approximately 10 min.

The patients were asked to fuldill a quality of life questionnaire (SF-36), which will be assessed in a future study regarding psychoacoustics for mechanical heart valve sounds.

Perspectives: The results obtained from this analysis will contribute to expand knowledge concerning the sound produced by these three different types of mechanical heart valve prosthesis. The study can add one important parameter in the choice of the implanted valve: patient's pleasantness. It will assess some of the most sold mechanical heart valve worldwide and the final results can contribute to elucidate which type, among those valves, that should be chosen to a specific patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age and older) with an aortic mechanical heart valve which belongs to one of the three investigated valve types and have been implanted from three months to four years before the investigation.

Exclusion Criteria:

* Patients with severe hearing impairment (evaluated by a conventional audiogram inside the sound-insulated chamber) or who use hearing aid;
* patients with severe cardiac arrhythmias;
* patients with claustrophobia;
* patients who are not capable of cooperating to the experimental conditions at a sound-insulated chamber;
* patients who are unable to fulfil the quality of life questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients are expected to be included. They all must have a mechanical heart valve in the aortic position implanted between 3 months and 4,5 years prior to the investigation. The patients will be divided into tree main groups, which correspond to the type of valve they have acquired - ATS (ATS Medical Inc, Minneapolis, MN, USA), Medtronic-Hall™ (Medtronic, Minneapolis, MN, USA) and St. Jude Medical Standard (St. Jude Medical Inc, St. Paul, MN, USA). With the purpose of recruiting a greater number of patients than those available in the geographic region of Denmark, we have established an agreement with The Heart Center in Bad Oeynhausen, Germany, who will contribute to the study with all 150 patients.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2005-11; Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thais A. Pedersen, doctor, Principal Investigator — University of Aarhus
Locations (1):
- Herz- und Diabeteszentrum Nordrhein Westfalen, Bad Oeynhausen, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 84 included patients were recruited from the same out patient clinic at the Heart Center, Bad Oeynhausen, Germany. They have been recruited between november 2005 and april 2006.
Pre-assignment Details: 3 previously included patients were excluded from the analysis due to double mechanical heart valve prosthesis (in both mitral and aortic position).
Groups:
- ATS (Open Pivot® Standard): patients with an ATS mechanical heart valve recruited from a cardiology outpatient clinic following heart valve replacement at the same hospital between three months and four years prior to this investigation.
- Medtronic Hall: patients with a Medtronic Hall mechanical heart valve recruited from a cardiology outpatient clinic following heart valve replacement at the same hospital between three months and four years prior to this investigation.
- St Jude Medical: patients with a St Jude Medical mechanical heart valve recruited from a cardiology outpatient clinic following heart valve replacement at the same hospital between three months and four years prior to this investigation.
Period: Overall Study
Arm/Group | ATS (Open Pivot® Standard) | Medtronic Hall | St Jude Medical
Started | 15 | 29 | 40
Completed | 15 | 29 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATS (Open Pivot® Standard) | Medtronic Hall | St Jude Medical | Total
Number analyzed (Participants) | 15 | 29 | 40 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0.0
  Between 18 and 65 years | 7 | 11 | 18 | 36.0
  >=65 years | 8 | 18 | 22 | 48.0
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (7) | 64 (9) | 63 (10) | 63 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 8 | 21.0
  Male | 8 | 23 | 32 | 63.0
Region of Enrollment [Number; unit: participants]
  Germany | 15 | 29 | 40 | 84.0

OUTCOME MEASURES:

1. Primary Outcome: Intensity (Highness) of the Sound From Mechanical Heart Valves
Description: The measurements took place in a Bioacoustic laboratory. The total background noise was 9 dB(A). The valve closing sounds were recorded by a microphone placed 5 cm above the patient's chest. This sound was pre-amplified, amplified, filtered and stored on an instrumentation recorder for later off-line analysis.
Time Frame: 10.06.2007
Population: Patients with a mechanical heart valve prosthesis recruited from a cardiology outpatient clinic following heart valve replacement at the same hospital between three months and four years prior to this investigation.
Measure: Mean (Standard Deviation); unit: dB (decibel)
Groups:
- Group 1 - ATS: patients with an ATS mechanical heart valve recruited from a cardiology outpatient clinic following heart valve replacement at the same hospital between three months and four years prior to this investigation.
- Group 2- Medtronic Hall: patients with a Medtronic Hall mechanical heart valve recruited from a cardiology outpatient clinic following heart valve replacement at the same hospital between three months and four years prior to this investigation.
- Group 3 - St Jude Medical: patients with a St Jude Medical mechanical heart valve recruited from a cardiology outpatient clinic following heart valve replacement at the same hospital between three months and four years prior to this investigation.
Arm/Group | Group 1 - ATS | Group 2- Medtronic Hall | Group 3 - St Jude Medical
Number analyzed (Participants) | 15 | 29 | 40
dB (decibel) | 43 (5) | 41 (4) | 40 (4)
Statistical Analysis 1: Comparison: Group 1 - ATS vs Group 2- Medtronic Hall vs Group 3 - St Jude Medical; The comparison of the three valve groups with respect to the objective sound measures was made by the one-way ANOVA method. The null hypothesis is that there is no difference on intensity of heart valve sounds among the three groups; Test type: Superiority or Other; p < 0.05, ANOVA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No